CLINICAL TRIAL: NCT03277066
Title: A 4-week, Randomized, Double-blind, Multicenter, Placebo-controlled Phase 2 Study to Evaluate the Efficacy and Safety of HP-5000 in Subjects With Osteoarthritis (OA) of the Knee
Brief Title: A 4-week Study to Evaluate the Efficacy and Safety of HP-5000 in Subjects With Knee Osteoarthritis
Acronym: HP-5000
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Noven Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Noven Therapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HP-5000-US-05
Record Dates: First submitted 2017-09-06; First posted 2017-09-08 (Actual); Results first posted 2021-12-23 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-11

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Diclofenac Sodium Active Topical Patch 1 (Experimental): Diclofenac sodium 1 topical patches will be compared against placebo patches.
  Interventions: Drug: Diclofenac Sodium Active Topical Patch 1; Drug: Placebo patch
- Diclofenac Sodium Active Topical Patch 2 (Experimental): Diclofenac sodium 2 topical patches will be compared against placebo patches.
  Interventions: Drug: Diclofenac Sodium Active Topical Patch 2; Drug: Placebo patch

INTERVENTIONS:
Drug: Diclofenac Sodium Active Topical Patch 1 — HP-5000 Active Topical Patch 1 were applied on subjects with Osteoarthritis of the knee(s)
  Other Names: HP-5000
  Arms: Diclofenac Sodium Active Topical Patch 1
Drug: Diclofenac Sodium Active Topical Patch 2 — HP-5000 Active Topical Patch 2 were applied on subjects with Osteoarthritis of the knee(s)
  Other Names: HP-5000
  Arms: Diclofenac Sodium Active Topical Patch 2
Drug: Placebo patch — Topical placebo patches were applied on subjects with Osteoarthritis of the knee(s)
  Other Names: Placebo treatment

SUMMARY:
A 4-week, Randomized, Double-blind, Multicenter, Placebo-controlled Phase 2 Study to Evaluate the Efficacy and Safety of HP-5000 in Subjects with Osteoarthritis (OA) of the Knee

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, and placebo-controlled phase 2 study evaluating 2 formulations of HP-5000 in subjects with OA of the knee. The study will consist of up to 28-day Screening Phase that will include a Washout Period of current prescription and over the counter (OTC) analgesics, a 4-week double-blind Treatment Phase, and a 1-week safety Follow-up Period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 40 to 85 years with a clinical diagnosis of OA of the target knee according to the American College of Rheumatology (ACR) criteria, including:
* Symptoms for at least 6 months prior to screening, AND
* Knee pain in the target knee for 30 days of the preceding month (periarticular knee pain due to OA and not due to other conditions such as bursitis, tendonitis, etc.) AND
* The pain in the target knee required the use of nonsteroidal anti-inflammatory drugs (NSAIDs) either over the counter (OTC) per recommendation of a physician or prescribed.

Exclusion Criteria:

* Body mass index (BMI) > 40
* Any subject who disobeyed the restriction of prohibited therapies (i.e., use rescue medication) during Screening Washout Period.
* Secondary OA of the knee (rheumatoid arthritis, gout, psoriasis, syphilitic neuropathy, ochronosis, metabolic or other primary bone disease or acute trauma).

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Klauss, MD, MSc, Study Director — Noven Pharmaceuticals, Inc.
Locations (1):
- Noven Pharmaceuticals, Inc., Jersey City, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Diclofenac Sodium Active Topical Patch 1: Diclofenac Sodium Active Topical Patch 1 and Diclofenac Sodium Active Topical Patch 2 contain the same amount of diclofenac sodium but in different formulations.
  Diclofenac Sodium Active Topical Patch 1 was applied to the target knee on subjects with Osteoarthritis of the knee(s) for 4-week treatment.
- Diclofenac Sodium Active Topical Patch 2: Diclofenac Sodium Active Topical Patch 1 and Diclofenac Sodium Active Topical Patch 2 contain the same amount of diclofenac sodium but in different formulations.
  Diclofenac Sodium Active Topical Patch 2 was applied to the target knee on subjects with Osteoarthritis of the knee(s) for 4-week treatment.
- Placebo Patch: Placebo patch was applied to the target knee on subjects with Osteoarthritis of the knee(s) for 4-week treatment.
Period: Overall Study
Arm/Group | Diclofenac Sodium Active Topical Patch 1 | Diclofenac Sodium Active Topical Patch 2 | Placebo Patch
Started | 71 | 72 | 146
Completed (These numbers are the Full Analysis Set population include all randomized subjects who have had at least 1 patch of double-blind study drug applied and who have at least 1 post-baseline assessment of the primary efficacy measure.) | 69 | 71 | 143
Not Completed | 2 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- HP-5000-75α Patch (5% Diclofenac Sodium): Diclofenac Sodium Active Topical Patch 1 and Diclofenac Sodium Active Topical Patch 2 contain the same amount of diclofenac sodium but in different formulations.
  Diclofenac Sodium Active Topical Patch 1 was applied to the target knee on subjects with Osteoarthritis of the knee(s for 4-week treatment.
- HP-5000-DRS400 Patch (5% Diclofenac Sodium): Diclofenac Sodium Active Topical Patch 1 and Diclofenac Sodium Active Topical Patch 2 contain the same amount of diclofenac sodium but in different formulations.
  Diclofenac Sodium Active Topical Patch 2 was applied to the target knee on subjects with Osteoarthritis of the knee(s) for 4-week treatment.
- Total: Total of all reporting groups
Arm/Group | HP-5000-75α Patch (5% Diclofenac Sodium) | HP-5000-DRS400 Patch (5% Diclofenac Sodium) | Placebo Patch | Total
Number analyzed (Participants) | 69 | 71 | 143 | 283
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 45 | 40 | 78 | 163
  >=65 years | 24 | 31 | 65 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (8.66) | 57.1 (8.65) | 59 (8.46) | 57.8 (8.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 36 | 73
  Male | 52 | 51 | 107 | 210
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 17 | 34 | 71
  Not Hispanic or Latino | 49 | 54 | 109 | 212
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 69 | 71 | 143 | 283
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.51 (5.103) | 29.83 (4.898) | 29.89 (5.257) | 29.78 (5.116)

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Efficacy & Safety of HP-5000 Topical Patches in Subjects With Osteoarthritis of the Knee: Change in Osteoarthritis Pain Score
Description: To evaluate efficacy of HP-5000 Active Topical Patch 1 and HP-5000 Active Topical Patch 2 compared with placebo for the treatment of Osteoarthritis of the knee as evaluated by change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain score from baseline to week 4. WOMAC pain score is a scale that evaluate five items including walking, stair climbing, nocturnal, rest and weight bearing. Each item is rated on a scale of 0 to 4, with 0 being no difficulty and 4 being extremely difficulty. The total score is the sum of five items. The total score range from 0 to 20 with a low score considered a better outcome and a high score considered a worse outcome.
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diclofenac Sodium Active Topical Patch 1 | Diclofenac Sodium Active Topical Patch 2 | Placebo Patch
Number analyzed (Participants) | 69 | 71 | 143
score on a scale | -6.3 (4.47) | -5.6 (4.06) | -5.2 (4.16)
Statistical Analysis 1: Comparison: Diclofenac Sodium Active Topical Patch 1 vs Placebo Patch; Test type: Superiority; p = 0.0110, Mixed Models Analysis; Lest-Squared Mean Differences = 0.0110
Statistical Analysis 2: Comparison: Diclofenac Sodium Active Topical Patch 2 vs Placebo Patch; Test type: Superiority; p = 0.2835, Mixed Models Analysis; Lest-Squared Mean Differences = 0.2835

2. Secondary Outcome: WOMAC Pain Score Week 2 Change From Baseline
Description: To evaluate efficacy of HP-5000 Active Topical Patch 1 and HP-5000 Active Topical Patch 2 compared with placebo for the treatment of Osteoarthritis of the knee as evaluated by change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain score from baseline to week 2. WOMAC pain score is a scale that evaluate five items including walking, stair climbing, nocturnal, rest and weight bearing. Each item is rated on a scale of 0 to 4, with 0 being no difficulty and 4 being extremely difficulty. The total score is the sum of five items. The total score range from 0 to 20 with a low score considered a better outcome and a high score considered a worse outcome. The total score range from 0 to 20 with a low score considered a better outcome and a high score considered a worse outcome.
Time Frame: Baseline and 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diclofenac Sodium Active Topical Patch 1 | Diclofenac Sodium Active Topical Patch 2 | Placebo Patch
Number analyzed (Participants) | 68 | 68 | 138
score on a scale | -5.8 (4.29) | -5.3 (3.67) | -5.0 (4.01)

3. Secondary Outcome: WOMAC Stiffness Score Change From Baseline
Description: To evaluate efficacy of HP-5000 Active Topical Patch 1 and HP-5000 Active Topical Patch 2 compared with placebo for the treatment of Osteoarthritis of the knee as evaluated by change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Score from baseline to week 4. The WOMAC Stiffness scale assesses 2 items including morning stiffness and stiffness occurring later in the day. Each item is rated on a scale of 0 to 4, with 0 being no difficulty and 4 being extremely difficulty. The total score is the sum of two items range from 0 to 8 with a low score considered as a better outcome.
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diclofenac Sodium Active Topical Patch 1 | Diclofenac Sodium Active Topical Patch 2 | Placebo Patch
Number analyzed (Participants) | 67 | 67 | 135
score on a scale | -2.4 (2.06) | -2.1 (1.94) | -1.7 (1.77)

4. Secondary Outcome: WOMAC Physical Function Score
Description: To evaluate efficacy of HP-5000 Active Topical Patch 1 and HP-5000 Active Topical Patch 2 compared with placebo for the treatment of Osteoarthritis of the knee as evaluated by change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) physical function score from baseline to week 4. The WOMAC Physical Function assesses the following 17 items using the 0 to 4 scale. These 17 items include: 1. descending stairs; 2. ascending stairs; 3. rising from sitting; 4. standing; 5. bending to floor; 6. walking on a flat surface; 7. getting in/getting out of car; 8. going shopping; 9. putting on socks; 10. lying in bed; 11. taking off socks; 12. rising from bed; 13. getting in/out of bath; 14. sitting; 15. getting on/off toilet; 16. heavy domestic duties; 17. light domestic duties. Each item is rated on a scale of 0 to 4, with 0 being no difficulty and 4 being extremely difficulty. Total score range from 0 to 68 with lower score considered a better outcome.
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diclofenac Sodium Active Topical Patch 1 | Diclofenac Sodium Active Topical Patch 2 | Placebo Patch
Number analyzed (Participants) | 69 | 71 | 143
score on a scale | -19.8 (14.85) | -19.3 (13.63) | -15.6 (13.07)

ADVERSE EVENTS:
Time Frame: 4 weeks
Groups:
- Diclofenac Sodium Active Topical Patch 2: Diclofenac Sodium Active Topical Patch 1 and Diclofenac Sodium Active Topical Patch 2 contain the same amount of diclofenac sodium but in different formulations.
  Diclofenac Sodium Active Topical Patch 1 was applied to the target knee on subjects with Osteoarthritis of the knee(s) for 4-week treatment.
Arm/Group | Diclofenac Sodium Active Topical Patch 1 | Diclofenac Sodium Active Topical Patch 2 | Placebo Patch
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/71 | 0/143
Serious Adverse Events (participants affected / at risk) | 0/69 | 1/71 | 1/143
Other Adverse Events (participants affected / at risk) | 9/69 | 8/71 | 19/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diclofenac Sodium Active Topical Patch 1 (N=69) | Diclofenac Sodium Active Topical Patch 2 (N=71) | Placebo Patch (N=143)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diclofenac Sodium Active Topical Patch 1 (N=69) | Diclofenac Sodium Active Topical Patch 2 (N=71) | Placebo Patch (N=143)
Product taste abnormal (General disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (3) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-10-31): https://cdn.clinicaltrials.gov/large-docs/66/NCT03277066/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-21): https://cdn.clinicaltrials.gov/large-docs/66/NCT03277066/SAP_001.pdf